CLINICAL TRIAL: NCT04990466
Title: A Phase IIb/3 Randomized, Multi-Center, Placebo-Controlled Noninferiority Study to Evaluate the Safety, Immunogenicity and Potential Efficacy of an rVSV-SARS-CoV-2-S Vaccine (IIBR-100) in Adults Compared to an Approved COVID-19 Vaccine
Brief Title: Phase 2b/3 Trial of VSV-ΔG SARS-CoV-2 Vaccine (BRILIFE) Against Approved Comparator Vaccine.
Acronym: BRILIFE002
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Production of the BriLife vaccine was halted by government sponsor
Sponsor: NeuroRx, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BriLife_001
Record Dates: First submitted 2021-08-03; First posted 2021-08-04 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: COVID-19
Keywords: COVID-19; SARS-CoV-2; Delta Variant; BRILIFE; VSV-ΔG
MeSH Terms: conditions — COVID-19 | interventions — rVSV-deltaG-spike COVID-19 vaccine

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, comparator-controlled non-inferiority trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All vaccinations will be prepared by a single, unblinded research pharmacist in a site removed from the clinical immunization site
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Vaccine (Experimental): IIBR-100 (VSV-ΔG) vaccine at 10 to the 8th strength in prime/boost separated by 28 days
  Interventions: Drug: IIBR-100
- Active Comparator (Active Comparator): A currently approved vaccine for COVID-19 administered in prime/boost separated by 28 days
  Interventions: Drug: Active Comparator

INTERVENTIONS:
Drug: IIBR-100 — Administration of IIBR-100 vaccine
  Arms: Active Vaccine
Drug: Active Comparator — Administration of a currently-approved vaccine for COVID-19
  Arms: Active Comparator

SUMMARY:
IIBR-100 (VSV-ΔG) is a self-propagating live virus vaccine that contains the spike protein of the Wuhan wild-type SARS-CoV-2 virus. Preclinical and phase 1/2 trials have demonstrated no safety signals of concern and have further demonstrated immunologic response that approximates the response seen in convalescent individuals. The purpose of this phase 2b/3 trial is to document the non-inferiority of IIBR-100 vs. an already-approved vaccine for COVID-19.

DETAILED DESCRIPTION:
STUDY RATIONALE:

The SARS-CoV-2 virus is responsible for the COVID-19 pandemic, perhaps the deadliest in 100 years. The pandemic emerged from Wuhan Province in China in December 2019 and was declared by the WHO Director-General a Public Health Emergency of International Concern on 30 January 2020. Early cases have been reported in Israel around February 2020, and at the time this protocol is being drafted. The virus has spread to 190 countries with more than 198 million confirmed cases and more than 4.2 million confirmed deaths as of August 2, 2021 (WHO website https://covid19.who.int/).

In an effort to curb the pandemic, the Israel Institute for Biological Research (IIBR) has developed a replication-competent recombinant VSVΔG-spike vaccine (rVSV-SARS-CoV-2-S, IIBR-100), in which the glycoprotein of VSV is replaced by the spike protein of the SARS-CoV-2 virus. Pre-clinical data suggested IIBR-100 as a safe, efficacious, and protective vaccine against SARS-CoV-2 infection. In addition, clinical experience from over 20,000 subjects vaccinated with Ervebo®, an Ebola vaccine developed by Merck & Co. and licensed by FDA in 2019, also supports the safety of the VSV-ΔG backbone. An overlapping Phase I/II study in Israel is showing a good safety profile. This study is intended to support late-stage clinical studies and eventual mass immunization of the Georgian population.

STUDY DESIGN:

This is a Phase IIb/3, prospective, randomized, comparator-controlled, observer-blind, multi-center non-inferiority study.

Subjects will receive two intramuscular (IM) injections of the IIBR-100 (prime-boost) separated by 28 days consisted of 1 ml replicating viral rVSV SARS-CoV-2-S vaccine or active comparator. Injection will be performed at Day 0 and Day 28±2d in the deltoid muscle and will be followed through 12 months post last vaccination.

Follow-up (FU) visits will occur 1, 2 and 4 weeks, as well as, 2 ,3, 6, 9, and 12 months post last vaccination.

The primary outcome will be PCR+ infection with COVID-19 six months after vaccination. Key secondary outcome will be serologic immunity.

Reactogenicity will be assessed at these visits, and blood will be drawn for immunogenicity assays. Additional safety and reactogenicity data will be solicited via electronic diary and telephone calls to subjects performed 1 and 2 days post each vaccination.

Reactogenicity will be measured by the occurrence of solicited injection site reaction and systemic reaction from the time of each vaccination through 7 days post each vaccination. Unsolicited non-serious Adverse Events (AEs), Serious adverse events (SAEs), new-onset chronic medical conditions (NOCMCs) and medically-attended adverse events (MAAEs) will be collected through 12 months after the last vaccination.

Clinical safety laboratory evaluations will be performed at screening, as well as immediately prior to and 7 days post each vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Males or females, ages 18 to 85 (inclusive) at the time of screening.
* Negative PCR and no presence of ELISA antibody titers to SARS-CoV-2 at screening.
* No clinically significant abnormalities in hematology, blood chemistry, or urinalysis laboratory tests at screening.
* Must agree not to enroll in another study of an investigational agent prior to completion of the study.
* Normal oral temperature, pulse rate no greater than 100 beats per minute (sinus rhythm) and controlled blood pressure (in the case of hypertensives under treatment, below 140/90 mmHg).
* Subjects must be able to understand the requirements of the study and must be accessible and willing to comply with the study procedures even under lock down conditions.
* Ability to provide informed consent -

Exclusion Criteria:

* History of severe local or systemic reactions to any vaccination or a history of severe allergic reactions or known allergy to the components of the vaccine, including allergy to rice.
* Receipt of investigational product (except of confirmed placebo in IIBR20-001 study) up to 30 days prior to screening or ongoing participation in another clinical trial (except of IIBR20-001 trial).
* Receipt of licensed vaccines within 14 days of planned study immunization and any AE's possibly related to licensed vaccine immunization at Day 0.
* Inability to observe possible local reactions at the injection sites due to a physical condition or permanent body art.
* Known hemoglobinopathy or coagulation abnormality (subjects treated by anticoagulation or anti platelets are not excluded).
* New onset of fever >37.8ºC AND [cough OR shortness of breath OR anosmia/ageusia], or any other inter current illness within 14 days prior to screening
* Factors that increase risk to the subject to severe disease per CDC guidance including the following risk factors (in any case of ambiguous grading, decision will be made per investigator's best clinical judgement): Cancer [ongoing malignancy or recently diagnosed malignancy in the last five years, not including non-melanotic skin cancer], Chronic Kidney Disease (eGFR<60 mL/min/1.73 m^2), liver disease (ALT or AST) > 1.5 × ULN; or alkaline phosphatase and direct bilirubin > ULN (total bilirubin may be up to 2 × ULN as long as direct bilirubin is equal to or below the ULN); or PT INR > 1.25), COPD; Immunocompromised state from solid organ transplant; Obesity (BMI≥30kg/m2); Serious heart conditions, such as heart failure, coronary artery disease, or cardiomyopathies; Sickle cell disease; Type 1/2 diabetes mellitus (HbA1C>8.0%, per medical history questioning or records) ); Asthma; Cerebrovascular disease; Cystic fibrosis, uncontrolled hypertension that does not respond to therapy, Pulmonary fibrosis, Thalassemia.

Anticipating the need for immunosuppressive treatment within the next 6 months. Clinically significant (by means of potentially risking the subject or that would be potentially detrimental to the results of the study) medical condition, physical examination findings, clinically significant abnormal laboratory results, or past medical history with clinically significant implications for current health or for severe COVID-19, per the investigator.

Any progressive or severe neurologic condition/disorder, dementia, seizure disorder, or history of Guillian-Barré syndrome.

* Known or suspected impairment of the immune system including rheumatic, connective tissue or vascular disease of autoimmune origin
* Clinically significant abnormal CBC results in WBC, hemoglobin, hematocrit, or platelets.
* Clinically significant abnormal urinalysis: RBC, protein, or glucose only.
* Positive serology for: hepatitis B surface antigen, hepatitis C, HIV.
* Known or suspected illness caused by coronaviruses, SARS-CoV 1, and Middle East Respiratory Syndrome (MERS)-CoV..
* Received any prior vaccine against a coronavirus.
* Receipt of blood/plasma products or immunoglobulin, from within 60 days before study intervention administration or planned receipt throughout the study.
* Immunosuppressive medications received within 90 days before screening. (Not including [1] corticosteroid nasal spray for allergic rhinitis; [2] topical corticosteroids for mild, uncomplicated dermatitis; or [3] oral/parenteral corticosteroids given for non-chronic conditions not expected to recur [length of therapy 10 days or less with completion at least 30 days prior to vaccination].)
* History of alcohol or drug abuse per clinical judgement within 5 years prior to study vaccination (excluding cannabis)
* Participants who, in the judgment of the investigator, will be unlikely to comply with the requirements of this protocol.
* Any other significant finding that in the opinion of the investigator would increase the risk of the individual having an adverse outcome from participating in this study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-09-30 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
Prevention of Serology-confirmed SARS-CoV-2 infection | 180 days
  Prevention of serology confirmed infection (seroconversion to non-vaccine antigen) in Prevention of PCR+ COVID-19 in combination with one or more of the clinical symptoms

SECONDARY OUTCOMES:
Prevention of COVID-19 mild/moderate disease | Beginning 14 days after second injection
  Prevention of COVID-19 mild/moderate disease
Prevention of COVID-19 severe disease | Beginning 14 days after second injection
  Prevention of COVID-19 severe disease
Serologic Immunogenicity | 365 days
  IIBR-100 Immunogenicity as determined by GMT, GMFR, Seroconversion rates of the neutralizing antibody titers to SARS-CoV-2 at baseline (day 0) and throughout the study
Cellular Immunogenicity | 365 days
  Cellular immunogenicity as assessed by ELISPOT and ELISA

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan C Javitt, MD, MPH, Study Chair — NRx Pharmaceuticals, Inc.

IPD SHARING:
Plan to Share IPD: Yes
Vaccination dates, baseline serology, and post-vaccination serology/cellular immunity/infection rates will be shared
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Protocol, SAP, and ICF will be shared prior to first patient visit. CSR will be shared following regulatory determination
Access Criteria: all qualified researchers